CLINICAL TRIAL: NCT03390608
Title: Prognosis, Prognostic Factors and Predictive Factors in Centimeter or Subcentimeter Node-negative Breast Cancer
Brief Title: Prognostic and Predictive Factors for Small Breast Tumors
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: The Swedish Society of Medicine (Other); The Swedish Breast Cancer Association (BRO) (Unknown); Swedish Breast Cancer Group (Other)
Responsible Party: Principal Investigator, Andreas Pettersson, Researcher, Principal Investigator, Karolinska Institutet
Other Study IDs: 365
Record Dates: First submitted 2017-12-15; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy; Trastuzumab; Drug Therapy; Receptors, Estrogen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women with T1ab breast cancer.
  Interventions: Drug: Endocrine therapy; Radiation: Radiotherapy; Drug: Herceptin; Drug: Chemotherapy; Procedure: Type of breast cancer surgery; Other: Age at diagnosis; Other: Screen detected tumor; Other: Menopausal status at diagnosis; Other: Tumor size; Other: Estrogen receptor (ER) status; Other: Tumor grade; Other: HER2-status; Other: Intrinsic subgroups of breast cancer; Other: Nodal status

INTERVENTIONS:
Drug: Endocrine therapy — Endocrine treatment versus no endocrine therapy (in women with hormone receptor positive1 disease).
Radiation: Radiotherapy — Radiotherapy versus no radiotherapy.
Drug: Herceptin — Trastuzumab versus no trastuzumab (in women with HER2-positive disease).
Drug: Chemotherapy — Chemotherapy versus no chemotherapy.
Procedure: Type of breast cancer surgery — Type of surgery (partial mastectomy, mastectomy, other).
Other: Age at diagnosis — Age at diagnosis (<35, 35-<50, 50-<70, ≥70).
Other: Screen detected tumor — Screening detected tumor (yes, no).
Other: Menopausal status at diagnosis — Menopausal status (premenopausal, postmenopausal).
Other: Tumor size — Tumor size (≤5 mm, 6-≤10 mm).
Other: Estrogen receptor (ER) status — ER-status (positive, negative).
Other: Tumor grade — Tumor grade (1, 2, 3).
Other: HER2-status — HER2-status (positive, negative).
Other: Intrinsic subgroups of breast cancer — Intrinsic subgroup proxy (Luminal A, Luminal B (HER2-negative), Luminal B (HER2-positive), HER2-positive (non-luminal), Triple negative).
Other: Nodal status — N-status (N0, N1).

SUMMARY:
Because of mammography screening increasingly more women are diagnosed with centimeter or subcentimeter node-negative breast cancer (i.e., T1abN0); these tumors account for approximately 19% of all newly diagnosed breast cancers in Sweden. Although the long term relapse-free survival rates among patients with such tumors is as high as ≥90%, some reports suggest that certain patient subgroups may have rates <75%. Firmly established prognostic and predictive factors for patients with T1abN0 tumors are, however, lacking. This is a nationwide, register-based cohort study investigating prognostic and predictive factors in women with centimeter or subcentimeter breast cancer. The study hypotheses are: 1) Established prognostic and/or predictive factors in overall breast cancer are prognostic and/or predictive factors also in centimeter or subcentimeter node-negative breast cancer; 2) The established relative reduction in risk of recurrence and death of adjuvant treatment for overall breast cancer are similar in centimeter or subcentimeter node-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female.
2. Operated for centimeter or subcentimeter breast cancer.

Exclusion Criteria:

1. Previous breast cancer.
2. Metastatic breast cancer at diagnosis.

Max Age: 100 Years | Sex: Female
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The study population consists of all Swedish women operated for centimeter or subcentimeter breast cancer who are included in the regional breast cancer registries (1977 to 2007) or the national breast cancer registry (2008 onwards).
Sampling Method: Non-Probability Sample
Enrollment: 35002 (Actual)
Dates: Start 1977-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2016-07-30 (Actual)

PRIMARY OUTCOMES:
Breast cancer specific death | January 1, 1977 to December 31, 2014

SECONDARY OUTCOMES:
Death from any cause | January 1, 1977 to July 30, 2016
Metachronous breast cancer | January 1, 1977 to July 30, 2016
  Ipsilateral or contralateral breast cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Instiutet, Solna, Sweden

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT03390608/SAP_000.pdf
  • Study Protocol (2014-02-22): https://cdn.clinicaltrials.gov/large-docs/08/NCT03390608/Prot_001.pdf